CLINICAL TRIAL: NCT06128512
Title: Evaluating the Efficacy of Auricular Acupuncture in Reducing Examination Anxiety Among Medical Students
Brief Title: Auricular Acupuncture Efficacy for Medical Students' Examination Anxiety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Medicine and Pharmacy at Ho Chi Minh City (Other)
Responsible Party: Principal Investigator, Bui Pham Minh Man, Investigator, University of Medicine and Pharmacy at Ho Chi Minh City
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 698/HDDD-DHYD
Record Dates: First submitted 2023-11-04; First posted 2023-11-13 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Anxiety; Anxiety, Exam
Keywords: anxiety; examination anxiety; acupuncture; auricular acupuncture; traditional medicine
MeSH Terms: conditions — Anxiety Disorders | interventions — Acupuncture, Ear

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participants will not know which group they are assigned to - either the intervention or placebo group. Sham auricular acupuncture (Sham-AA) will be administered similarly to AA but without the use of needles.
  The physician administering the treatments will be aware of the group assignments but will not be involved in result assessment or data analysis. Those responsible for outcome evaluation and data analysis will not know the treatment allocations.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AA (Experimental): Auricular acupuncture (AA) 24 hours before the examination.
  Interventions: Other: Auricular acupuncture
- Sham-AA (Sham Comparator): Sham Auricular acupuncture (Sham-AA) 24 hours before the examination.
  Interventions: Other: Sham Auricular acupuncture

INTERVENTIONS:
Other: Auricular acupuncture — Auricular acupuncture is administered 24 hours before the examination using patches, each possessing a square shape with a side length of 10 mm, coupled with a sterilized needle measuring 0.25 x 1.3 mm. Four acupoints are selected on one ear, including the Master cerebral point, Tranquilizer point, Relaxation point, and Heart point (CO15). The patch containing the needle will remain in place until the student completes the examination.
  Arms: AA
Other: Sham Auricular acupuncture — Sham Auricular acupuncture is administered 24 hours before the examination using patches, each possessing a square shape with a side length of 10 mm, without a needle. Four acupoints are selected on one ear, including the Master cerebral point, Tranquilizer point, Relaxation point, and Heart point (CO15). The patch will remain in place until the student completes the examination.
  Arms: Sham-AA

SUMMARY:
Anxiety is a natural human response when facing challenging circumstances or threats to oneself. It is highly prevalent, estimated to range from 3.8% to 25%. Anxiety significantly impacts daily life and the overall quality of life. Of particular concern is the potential for anxiety to increase cardiovascular risk factors such as hypertension, a higher incidence of heart disease, and premature mortality.

Anxiety occurs in nearly everyone, but university students are particularly prone to experiencing anxiety and higher levels of mental stress compared to the general population. This trend is notably pronounced among medical students, a group with a significantly higher prevalence of anxiety that can reach as high as 90%. Multiple factors contribute to this anxiety and stress, notably the pressure of academic examinations.

Several studies suggest that acupuncture not only positively affects anxiety but also has fewer side effects compared to pharmacological treatments. Among these, a form of acupuncture known as auricular acupuncture (AA) is considered safe and has demonstrated effectiveness in reducing pre-surgical and dental anxiety. However, evidence supporting its effectiveness in reducing examination anxiety among medical students remains insufficient. Hence, in this study, we have designed a randomized controlled trial, including a placebo arm, to establish the efficacy and safety of AA in addressing this issue.

DETAILED DESCRIPTION:
Medical students with examination anxiety, identified by a score equal to 40 or more on the STAI-Y1 scale, will be selected and randomly allocated into two groups: the intervention group (AA group) and the placebo group (Sham-AA), at a 1:1 allocation ratio.

The intervention will be carried out 24 hours before the examination and will be monitored until the students complete the test. In the AA group, AA devices will be utilized, while adhesive patches without needles will be used in the Sham-AA group.

Data regarding anxiety levels will be recorded through scores obtained from the STAI-Y1 questionnaire and VAS-100; heart rate, diastolic blood pressure, systolic blood pressure, examination scores, and adverse events will also be evaluated at various intervals.

ELIGIBILITY:
Inclusion Criteria:

* Medical students preparing to take an examination for a course experience anxiety with a STAI-Y1 score of 40 or higher.
* Voluntary informed consent.

Exclusion Criteria:

* Currently experiencing additional anxiety alongside the impending examination anxiety.
* Using stimulants within 24 hours prior.
* Recent use of any drugs impacting intervention outcomes including psychotropic medications, blood pressure, and heart rate-affecting medications.
* History of alcohol or substance addiction.
* History of cardiac and neuropsychiatric disorders.
* Prior experience with auricular acupuncture.
* History of hypersensitivity reactions to any form of acupuncture with needles.
* Existing injuries or lesions at the acupoints being investigated in this study.
* Presence of severe medical conditions (e.g., cardiovascular, hepatic, renal, or others) that could potentially influence treatment outcomes as assessed by researchers.
* Currently enrolled in another intervention study.
* Pregnancy or lactating.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2023-11-15 (Actual); Primary Completion 2024-03-27 (Actual); Study Completion 2024-04-28 (Actual)

PRIMARY OUTCOMES:
Changes in the State-Trait Anxiety Inventory Form Y1 (STAI-Y1) score | immediately pre-intervention (T0), 30 minutes (T1), 24 hours (T2)
  The STAI-Y1 comprises 20 questions, each rated on a 4-point scale from 1 "not at all" to 4 "very much so". Therefore, the STAI-Y1 score ranges from 20 to 80, with higher scores indicating increased levels of anxiety.

SECONDARY OUTCOMES:
Changes in Visual Analog Scale (VAS) score for anxiety | immediately pre-intervention (T0), 30 minutes (T1), 24 hours (T2)
  The VAS includes a 100mm line with endpoints labeled from "no anxiety" to "greatest anxiety ever experienced". Participants will mark on the line the point that represents their current level of anxiety. The VAS score ranges from 0 to 100, with higher scores indicating increased levels of anxiety.
Changes in Diastolic Blood Pressure | immediately pre-intervention (T0), 30 minutes (T1), 24 hours (T2)
  Diastolic blood pressure is measured using an electronic device, in units of mmHg, conducted by investigators. The higher the value, the higher the diastolic blood pressure.
Changes in Systolic Blood Pressure | immediately pre-intervention (T0), 30 minutes (T1), 24 hours (T2)
  Systolic blood pressure is measured using an electronic device, in units of mmHg, conducted by investigators. The higher the value, the higher the systolic blood pressure.
Changes in heart rate | immediately pre-intervention (T0), 30 minutes (T1), 24 hours (T2)
  Heart rate is measured using an electronic device, in units of beats per minute, conducted by investigators. The higher the value, the faster the heart rate.
The examination score | up to 1 month
  The examination scores will be recorded after the students receive their test results. The scoring scale ranges from 0 to 10 points. Higher scores indicate a better performance on the examination.
Proportion of intervention-related adverse effects | during the intervention
  Anticipated adverse events (AEs) from auricular acupuncture (AA) may comprise pain at the insertion site, local discomfort, skin irritation (itching and redness), inflammation, bleeding, chondritis, dizziness, nausea, and hypersensitivity reactions.
  Moreover, any unanticipated AEs related to AA will be recorded and observed.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Traditional medicine, University of Medicine and Pharmacy at Ho Chi Minh City, Ho Chi Minh City, Vietnam

REFERENCES:
- [Background] Remes O, Brayne C, van der Linde R, Lafortune L. A systematic review of reviews on the prevalence of anxiety disorders in adult populations. Brain Behav. 2016 Jun 5;6(7):e00497. doi: 10.1002/brb3.497. eCollection 2016 Jul. PMID 27458547
- [Background] Roest AM, Martens EJ, de Jonge P, Denollet J. Anxiety and risk of incident coronary heart disease: a meta-analysis. J Am Coll Cardiol. 2010 Jun 29;56(1):38-46. doi: 10.1016/j.jacc.2010.03.034. PMID 20620715
- [Background] Mboya IB, John B, Kibopile ES, Mhando L, George J, Ngocho JS. Factors associated with mental distress among undergraduate students in northern Tanzania. BMC Psychiatry. 2020 Jan 29;20(1):28. doi: 10.1186/s12888-020-2448-1. PMID 31996200
- [Background] Fares J, Al Tabosh H, Saadeddin Z, El Mouhayyar C, Aridi H. Stress, Burnout and Coping Strategies in Preclinical Medical Students. N Am J Med Sci. 2016 Feb;8(2):75-81. doi: 10.4103/1947-2714.177299. PMID 27042604
- [Background] Li M, Li WQ, Li LMW. Sensitive Periods of Moving on Mental Health and Academic Performance Among University Students. Front Psychol. 2019 Jun 13;10:1289. doi: 10.3389/fpsyg.2019.01289. eCollection 2019. PMID 31263436
- [Background] Bae H, Bae H, Min BI, Cho S. Efficacy of acupuncture in reducing preoperative anxiety: a meta-analysis. Evid Based Complement Alternat Med. 2014;2014:850367. doi: 10.1155/2014/850367. Epub 2014 Sep 2. PMID 25254059
- [Background] Amorim D, Amado J, Brito I, Fiuza SM, Amorim N, Costeira C, Machado J. Acupuncture and electroacupuncture for anxiety disorders: A systematic review of the clinical research. Complement Ther Clin Pract. 2018 May;31:31-37. doi: 10.1016/j.ctcp.2018.01.008. Epub 2018 Jan 31. PMID 29705474
- [Background] Karst M, Winterhalter M, Munte S, Francki B, Hondronikos A, Eckardt A, Hoy L, Buhck H, Bernateck M, Fink M. Auricular acupuncture for dental anxiety: a randomized controlled trial. Anesth Analg. 2007 Feb;104(2):295-300. doi: 10.1213/01.ane.0000242531.12722.fd. PMID 17242083
- [Background] Zanella S, Buccelletti F, Vassiliadis A, De Bortoli R, Visentini S, Pedrotti G, Azzalin L. Preoperative anxiety management: acupuncture vs. pharmacological treatment - A prospective study. Eur Rev Med Pharmacol Sci. 2022 Feb;26(3):900-905. doi: 10.26355/eurrev_202202_27999. PMID 35179756
- [Background] Michalek-Sauberer A, Gusenleitner E, Gleiss A, Tepper G, Deusch E. Auricular acupuncture effectively reduces state anxiety before dental treatment--a randomised controlled trial. Clin Oral Investig. 2012 Dec;16(6):1517-22. doi: 10.1007/s00784-011-0662-4. Epub 2012 Jan 6. PMID 22219023
- [Background] Wang SM, Peloquin C, Kain ZN. The use of auricular acupuncture to reduce preoperative anxiety. Anesth Analg. 2001 Nov;93(5):1178-80, table of contents. doi: 10.1097/00000539-200111000-00024. PMID 11682391
- [Background] Favre-Felix J, Laurent V, Branche P, Huissoud C, Raffin M, Pradat P, Aubrun F, Dziadzko M. Auricular Acupuncture for Preoperative Anxiety in Parturient Women with Scheduled Cesarean Section: A Randomized Placebo-Controlled Blind Study. J Integr Complement Med. 2022 Jul;28(7):569-578. doi: 10.1089/jicm.2021.0346. Epub 2022 Apr 8. PMID 35394895